CLINICAL TRIAL: NCT02693093
Title: A Phase 1, Single Dose PK and Safety Study With NI-03 Followed by a Phase 2, Randomized, Double-Blind, Parallel-Group Dose-Ranging Study to Evaluate the Safety and Efficacy of NI-03 When Compared to Placebo in Subjects With Chronic Pancreatitis
Brief Title: A Dose Ranging Study Evaluating Efficacy and Safety of NI-03
Acronym: Tactic
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kangen Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NI03-001
Record Dates: First submitted 2016-02-12; First posted 2016-02-26 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): TID Day for 28 Days
  Interventions: Drug: Placebo
- 100 mg NI-03 (Experimental): TID Day for 28 Days
  Interventions: Drug: NI-03
- 200 mg NI-03 (Experimental): TID Day for 28 Days
  Interventions: Drug: NI-03
- 300 mg NI-03 (Experimental): TID Day for 28 Days
  Interventions: Drug: NI-03

INTERVENTIONS:
Drug: NI-03
  Arms: 100 mg NI-03; 200 mg NI-03; 300 mg NI-03
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of NI-03.

DETAILED DESCRIPTION:
The primary objective of the Single-Dose Phase is to assess the pharmacokinetics (PK) and safety of single doses of NI-03 when administered at doses of 100 mg, 200 mg or 300 mg to subjects with chronic pancreatitis.

The primary objective of the Double-Blind Phase of the study is to determine the efficacy, PK and safety of three doses of NI-03 (100 mg, 200 mg and 300 mg) as compared to placebo when administered three times daily (TID) for 28 consecutive days in subjects with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, subjects must meet all of the following criteria at Screening:

1. Males and females aged 18 to 85 years, inclusive, at the time of consent
2. Ability to communicate effectively with clinic site staff, ability and willingness to comply with the study schedule, restrictions, and requirements
3. Institutional Review Board (IRB)-approved written informed consent
4. Diagnosis of chronic pancreatitis
5. Baseline average daily worst pain score must be a minimum of 4 using the Numeric Rating Scale (NRS) during the 7-day run-in period
6. Patients on a non-opioid analgesic regimen that is expected to remain stable during the study period, or an opioid regimen with a morphine-equivalent dose not more than 100 mg daily.

Exclusion Criteria:

To be eligible to participate in this study, subjects must not meet any of the following criteria:

1. Any other clinically significant medical condition
2. Treatment with any investigational product within 14 days of Day 1 (or 5 drug half-lives if 5 drug half-lives are expected to exceed 14 days) of Day -7
3. Major abdominal surgery within 90 days of Day 1
4. History or presence of clinically significant cardiovascular disease
5. History of any cancer, except non-melanoma skin cancer, within 5 years of study enrollment,
6. History of endoscopic intervention within the previous 3 months or presence of a pancreatic duct stent
7. History of illicit drug abuse (i.e. use of any 'illegal' drugs within 6 months)
8. Active heavy alcohol use (defined as more than 2 alcoholic drinks per day or 14 alcoholic drinks per week)
9. Inadequate venous access
10. Significant blood loss, donation of ≥450 mL of blood, or blood or blood product transfusion within 7 days of Day 1
11. History or presence of hepatitis B (surface antigen positivity), active hepatitis C or human immunodeficiency virus (HIV) antibody
12. Active infection within 30 days of Day 1
13. Pregnant, planning to become pregnant or breast feeding
14. Positive urine or serum pregnancy test result at Screening or on Day 1
15. Active major psychiatric illness requiring a change in treatment within 3 months that would confound pain assessments
16. History of seizures within the last 12 months
17. Current use of anticonvulsants, antipsychotics, systemic steroids and, immunosuppressant therapy. *Use of gabapentin, pregabalin and benzodiazepines as treatment for chronic pancreatitis pain are allowed.
18. Presence of generalized pain syndrome apart from chronic pancreatitis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose
  Pharmacokinetic (PK) parameters such as Maximum concentration (Cmax), time to maximum concentration (Tmax), minimum concentration(Cmin), area under the curve (AUC), half-life (t1/2), apparent clearance (CL/F), and apparent volume of distribution (Vz/F) are assessed.
Phase 1 - Safety and Tolerability - Treatment Emergent Adverse Events (TEAE) via CTCAE v4.0 | through 7 days post-dose
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Phase 1 - Safety and Tolerability - Laboratory test results | through 7 days post-dose
  Laboratory test results will be graded and summarized based on CTCAE v4.03. and by shifts in results before and after dosing
Phase 2 - Efficacy Analysis - average daily worst pain intensity score | 4 Weeks

SECONDARY OUTCOMES:
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA -area under the curve (AUC) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA - Maximum concentration (Cmax) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA - time to maximum plasma concentration (tmax) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA - apparent clearance (CL/F) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA - plasma terminal half-life (t1/2) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 1 - To determine the pharmacokinetic profile for FOY251 and GBA - apparent volume of distribution (Vz/F) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 2 - Efficacy Analysis - Change from baseline in least pain score | change from baseline to Week 4
Phase 2 - Efficacy Analysis - Change from baseline in average pain score | 4 Weeks
Phase 2 - Efficacy Analysis - Change from baseline in current pain score | 4 Weeks
Phase 2 - Efficacy Analysis - Change from baseline in average morphine-equivalent daily opioid daily dose | 4 Weeks
Phase 2 - Efficacy Analysis - Change from baseline in quality of life | change from baseline to Week 4
  assessed using the pain interference aspects of the Brief Pain Inventory (BPI)
Phase 2 - Safety and Tolerability - Treatment Emergent Adverse Events (TEAE) via CTCAE v4.0 | Through day 57 (End of Study Visit)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Phase 2 - Safety and tolerability - Laboratory Test Results | Through day 57 (End of Study Visit)
  Laboratory test results will be graded and summarized based on CTCAE v4.03. and by shifts in results before and after dosing
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA -area under the curve (AUC) | Days 1 and 29, and at 0.25, 0.5, 1, 2 and 4 hours post-dose
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA - Maximum concentration (Cmax) | pre-dose and at 0.25, 0.5, 1, 2, 4 and 8 hours post-dose.
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA - time to maximum plasma concentration (tmax) | Days 1 and 29, and at 0.25, 0.5, 1, 2 and 4 hours post-dose
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA - plasma terminal half-life (t1/2) | Days 1 and 29, and at 0.25, 0.5, 1, 2 and 4 hours post-dose
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA - apparent clearance (CL/F) | Days 1 and 29, and at 0.25, 0.5, 1, 2 and 4 hours post-dose
Phase 2 - To determine the pharmacokinetic profile for FOY251 and GBA - apparent volume of distribution (Vz/F) | Days 1 and 29, and at 0.25, 0.5, 1, 2 and 4 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Phiip Hart, MD, Principal Investigator — OSU
Locations (48):
- United States (28):
  - University of Arkansas, Little Rock, Arkansas
  - Kaiser Permanente Medical Group, Los Angeles, California
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado-Div of Gastroenterology and Hepatology, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida - Division of Gastroenterology, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - The Carle Foundation Hospital, Urbana, Illinois
  - Indiana University - Indiana University Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University School of Medicine, New York, New York
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University (OSU) - Wexner Medical Center, Columbus, Ohio
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Texas Clinical Research Institute, Arlington, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Mason, Seattle, Washington
  - Wisconsin Center for Advanced Research, a division of GI Associates LLC, Milwaukee, Wisconsin
- Russia (8):
  - Federal Research Centre Institute of Cytology and Genetics, Novosibirsk
  - Military Medical Academu, Dep of Therapy of Adv. Training, Saint Petersburg
  - Military Medical Academy, Department of Hospital Therapy, Saint Petersburg
  - 1st Saint Petersburg State Medical University, Saint Petersburg
  - City Hospital #40, Saint Petersburg
  - City Polyclinic #4, Saint Petersburg
  - Medical University "Reaviz", Samara
  - Tomsk Regional Clinical Hospital, Tomsk
- Ukraine (12):
  - Institute of Gastroenterology, Dnipro
  - Central city Clinical Hospital, Therapeutic Department #2, Ivano-Frankivsk
  - Malaya Therapy National Institute, Kharkiv
  - City Policlinic #9, Kharkiv
  - City Hospital Named After Tropins, Therapy Department #1, Kherson
  - OK Clinic, Kyiv
  - Medical Center "Consilium Medical", Kyiv
  - Emergency Care Hospital, #1 Therapeutic Department, Lviv
  - Regional Hospital, Department of General Surgery, Odesa
  - 1st City Clinical Hospital, Therapeutic Department, Poltava
  - City Clinical Hospital #1, Gastroenterology Department, Vinnytsia
  - Medical Centre Diaservis, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hart PA, Osypchuk Y, Hovbakh I, Shah RJ, Nieto J, Cote GA, Avgaitis S, Kremzer O, Buxbaum J, Inamdar S, Fass R, Phillips RW, Yadav D, Ladd AM, Al-Assi MT, Gardner T, Conwell DL, Irani S, Sheikh A, Nuttall J; TACTIC Study Investigators. A Randomized Controlled Phase 2 Dose-Finding Trial to Evaluate the Efficacy and Safety of Camostat in the Treatment of Painful Chronic Pancreatitis: The TACTIC Study. Gastroenterology. 2024 Apr;166(4):658-666.e6. doi: 10.1053/j.gastro.2023.12.008. Epub 2023 Dec 15. PMID 38103842
- [Derived] Ramsey ML, Nuttall J, Hart PA; TACTIC Investigative Team. A phase 1/2 trial to evaluate the pharmacokinetics, safety, and efficacy of NI-03 in patients with chronic pancreatitis: study protocol for a randomized controlled trial on the assessment of camostat treatment in chronic pancreatitis (TACTIC). Trials. 2019 Aug 14;20(1):501. doi: 10.1186/s13063-019-3606-y. PMID 31412955